CLINICAL TRIAL: NCT02344706
Title: Diagnostic Value of Prehospital EEG in Non-convulsive Status Epilepticus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Johannes Björkman, Resident, Helsinki University Central Hospital
Other Study IDs: 237/3 03.12.2012
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy; Status Epilepticus
Keywords: Emergency Care, Prehospital; Coma; Electroencephalography
MeSH Terms: conditions — Epilepsy; Status Epilepticus; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mini-EEG, NCSE: Unconscious patients due to seizures, of whom EEG is registered
  Interventions: Device: Registration of EEG

INTERVENTIONS:
Device: Registration of EEG — EEG is registered for study purposes. No interventions to patient care is done at this stage. Acquisition is done without harming the patient.

SUMMARY:
A large proportion of patients (up to 20%) who suffer from an epileptic seizure and remain unconscious suffer from a non-convulsive epileptic seizure. The condition is difficult to diagnose, and impossible without the required instruments. Electroencephalogram is required in the diagnosis of non-convulsive status epilepticus. Presently, the diagnostic value and implementation of such a device in the prehospital field is little studied. The aim of this study is to evaluate the diagnostic value of the acquired electroencephalogram with a prototype EEG/EKG adapter connected to a Physio-Control LifePak 15 defibrillator/monitor. The EEG is registered in a otherwise normal fashion with scalp-electrodes, but only three channels are monitored, as this is deemed sufficient for the prehospital field, as well as for monitoring the epileptic seizures.

ELIGIBILITY:
Inclusion Criteria:

* Unconsciousness due to seizures in the prehospital field

Exclusion Criteria:

* Cardiac arrest
* Traumatic unconsciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients unconscious due to seizures in the prehospital field
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of EEG | 60min
  EEG signal assessed by a physician educated in interpretation of EEG, use a numeric scale (eg 0=not of value/corrupted, 5=good signal with diagnostic value)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Silfvast, MD, Phd, Study Director — Helsinki University Central Hospital; Johannes Björkman, MD, Principal Investigator — Helsinki University Central Hospital; Salmi Tapani, MD, PHD, Study Director — Helsinki University Central Hospital